CLINICAL TRIAL: NCT06398938
Title: EROS 3 Study Evaluation of Ultraaccelerated High Dose Rate Intrauterine Interventional Radiotherapy Brachytherapy in Terms of Overall Toxicity and Sexual Activity
Brief Title: Evaluation of Ultraaccelerated High Dose Rate Intrauterine Interventional Radiotherapy
Acronym: EROS3
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 6676
Record Dates: First submitted 2024-04-24; First posted 2024-05-03 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Locally Advanced Cervical Carcinoma
Keywords: cervical carcinoma; interventional radiotherapy; acute and late toxicities; radiochemotherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Interventional Radiotherapy — The patients will undergo four IRT fractions in one week

SUMMARY:
To evaluate the degree of acute and long-term intestinal, urinary and vaginal toxicity, and the impact on sexual activity of an accelerated fractionation of high dose rate interventional radiotherapy (IRT-HDR) in patients with locally advanced cervical cancer (IB2 - VA, N+/-).

DETAILED DESCRIPTION:
Observational, monocentric and prospective study. All patients with locally advanced cervix cancer will be underwent to radiochemotherapy followed by accelerated interventional radiotherapy (brachytherapy). Fist endpoints wer severe acute and late gastrointestinal, and urinary toxicities and sexual activity.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* ECOG 0-2
* Histological diagnosis of squamous carcinoma and/or adenocarcinoma of the uterine cervix
* FIGO IB2 Stadium - IVA (staging 20018)
* No contraindications to performing MRI of the pelvis
* Informed consent

Exclusion Criteria:

* Age <18 years
* PS >2
* Previous cancer in the last 10 years
* Previous radiation treatment in the region of interest
* Presence of pathologies that contraindicate radiotherapy treatment (genetic syndromes of hyper-radiosensitivity, ulcerative colitis, diverticulitis in the acute phase, severe diverticulosis, chronic pelvic inflammation)
* Presence of internal diseases that contraindicate chemotherapy or radio-chemotherapy treatment (severe liver disease, heart disease, renal failure, etc.)
* Presence of distant metastases in sites other than the pelvic lymph nodes
* Any significant medical condition that in the opinion of the investigator may interfere with the patient's optimal participation in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with locally advanced cervix cancer
Sampling Method: Non-Probability Sample
Enrollment: 129 (Estimated)
Dates: Start 2024-05-06 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Acute and late gastrointestinal toxicity | 6 months
  Acute and late toxicities will evaluated with CTCAE scale to analyze the safety of accelerated interventional radiotherapy
Acute and late urinary toxicity | 6 months
  Acute and late urinary toxicities will evaluated with CTCAE scale to analyze the safety of accelerated interventional radiotherapy
Sexual activity | 6 months
  Sexual activity will evaluated with CTCAE scale to analyze the safety of accelerated interventional radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: VALENTINA LANCELLOTTA, Principal Investigator — Fondazione Universiataria Policlinico A Gemelli IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli, IRCCS, Rome, Italy